CLINICAL TRIAL: NCT00007709
Title: CSP #706D - HIV Seroprevalence and Risks in Veterans With Severe Mental Illness
Brief Title: To Determine the Prevalence of HIV and Other Related Infections Such as Hepatitis C, Along With Associated Risk Behaviors, in Patients With Severe Mental Illness (SMI).
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Butterfield, Marian - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 706D
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Hepatitis C; HIV Infections; Mental Disorders
Keywords: Hepatitis C; HIV; severe mental illness (SMI)
MeSH Terms: conditions — Hepatitis C; HIV Infections; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
It is suspected, but not well documented, that persons with severe mental illness (SMI) represent a significant transmission source of serious infectious diseases. SMI diagnoses are defined as schizophrenia, schizoaffective disorder, bipolar disorder, or posttraumatic stress disorder (PTSD). Severely mentally ill persons are at high risk for Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome (HIV/AIDS). To assess the risk of HIV and related infections among these individuals, the National Institute of Mental Health (NIMH) Office on AIDS funded the HIV/SMI five site collaborative study "Assessing HIV/AIDS and Associated Health Risks in People with Severe Mental Illness". This Durham ERIC study supplements the NIMH HIV/SMI study with a four-year longitudinal cohort study of 300-plus SMI veterans in order to estimate the prevalence of HIV risk behaviors and HIV infection, as well as to measure utilization of health services over time. The Durham VA is the only VA site represented in the study and is collaborating with four non-VA sites including Dartmouth, University of New Hampshire, University of Connecticut and Duke University. As such, we have the additional goals of investigating health and health-care-service issues relevant to veterans with SMI and of establishing a database for the longitudinal study of veterans with SMI.

DETAILED DESCRIPTION:
Primary Objectives: To determine the prevalence of HIV and other related infections such as Hepatitis C, along with associated risk behaviors, in patients with severe mental illness (SMI).

Secondary Objectives: To identify the implications for mental health and medical services and to obtain a better understanding of the contextual factors that affect the health problems associated with HIV risk behavior.

Primary Outcomes: The primary outcome variables are HIV seroprevalence, prevalence of HIV risk behaviors including injection drug use and sexual promiscuity, personal and social-contextual factors, comorbid mental disorders, and health service use among SMI persons in each group, veterans versus non-veterans.

Intervention: N/A

Study Abstract: It is suspected, but not well documented, that persons with severe mental illness represent a significant transmission source of serious infectious diseases. SMI diagnoses are defined as schizophrenia, schizoaffective disorder, bipolar disorder, or posttraumatic stress disorder (PTSD). Severely mentally ill persons are at high risk for Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome (HIV/AIDS). To assess the risk of HIV and related infections among these individuals, the National Institute of Mental Health (NIMH) Office on AIDS funded the HIV/SMI five site collaborative study "Assessing HIV/AIDS and Associated Health Risks in People with Severe Mental Illness". This Durham ERIC study supplements the NIMH HIV/SMI study with a four-year longitudinal cohort study of 300-plus SMI veterans in order to estimate the prevalence of HIV risk behaviors and HIV infection, as well as to measure utilization of health services over time. The Durham VA is the only VA site represented in the study and is collaborating with four non-VA sites including Dartmouth, University of New Hampshire, University of Connecticut and Duke University. As such, we have the additional goals of investigating health and health-care-service issues relevant to veterans with SMI and of establishing a database for the longitudinal study of veterans with SMI.

Study participation consisted of a one-hour structured HIV-risk behavior interview and a blood and urine sample. These samples are being tested for HIV, syphilis, hepatitis B and C, cytomegalovirus, gonorrhea, and chlamydia at the Durham VA Microbiology Laboratory. Subject enrollment for this study concluded 6/30/2000 with 399 total subjects enrolled. Of these 399 enrolled, 111 subjects were re-tested and re-interviewed. The percentage of subjects enrolled at the Durham VAMC with infectious diseases is as follows: 2.6% with HIV infection; 21% with Hepatitis B core antibodies; and, 18% with Hepatitis C antibodies. Clinical management of subjects with positive serology continues to be administered according to the procedures developed by Richard Frothingham, M.D.

Final Results: The initial manuscript for the study was published in American Journal of Public Health in January, 2001 and analyses for additional publications are underway. Final Report to be submitted to Durham ERIC within 90 days of study end date (3/31/02).

ELIGIBILITY:
Inclusion Criteria:

SMI veterans

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-01

CONTACTS AND LOCATIONS:
Overall Officials: Marian I. Butterfield, MD MPH, Study Chair — VA Medical Center
Locations (1):
- VA Medical Center, Durham, North Carolina, United States